CLINICAL TRIAL: NCT04890678
Title: The Use of a Fully Automated Pulsating Support System (CuroCell® A4 CX20) in Pressure Ulcer Prevention and Treatment: a Clinical Test in 10 Belgian Nursing Homes
Brief Title: The Use of a Fully Automated Pulsating Support System (CuroCell® A4 CX20) in Pressure Ulcer Prevention and Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Care of Sweden AB (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EC/2018/1291
Record Dates: First submitted 2021-05-05; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2019-10

CONDITIONS: Pressure Ulcer; Pressure Injury; Pressure Sore; Pressure Ulcer, Buttock
Keywords: support surface; Elderly; Nursing home; prevention; treatment
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 22 residentsat risk for PU development (Experimental): 22 residents at risk for PU development, defined by a Braden score < 12 and/or a Braden subscale 'Mobility' score ≤ 2 and/or the presence of non-blanchable erythema in the sacral area.
  aged 65 years or over
  Interventions: Device: 22 residentsat risk for PU development
- 18 residents at least one PU category III-IV in the sacral area (Experimental): 18 residents at least one PU category III-IV in the sacral area aged 65 years or over
  Interventions: Device: 18 residents at least one PU category III-IV in the sacral area

INTERVENTIONS:
Device: 22 residentsat risk for PU development — mattress in bed
  The presence of PUs will be evaluated using the European Pressure Ulcer Advisory Panel (EPUAP) classification system (NPUAP, 2014) and the presence of incontinence- associated dermatitis (IAD) will be categorized using the Ghent Global IAD Categorisation Tool (GLOBIAD). For each participant, the Patient Repositioning Tool Ghent (PROTECT) will be used to individually recommend the frequency of skin observations and the frequency of repositioning.
  Arms: 22 residentsat risk for PU development
Device: 18 residents at least one PU category III-IV in the sacral area — mattress in bed The presence of PUs will be evaluated using the European Pressure Ulcer Advisory Panel (EPUAP) classification system (NPUAP, 2014) and the presence of incontinence- associated dermatitis (IAD) will be categorized using the Ghent Global IAD Categorisation Tool (GLOBIAD). For each participant, the Patient Repositioning Tool Ghent (PROTECT) will be used to individually recommend the frequency of skin observations and the frequency of repositioning.
  In the group of participants with a PU category III or IV, the Pressure Ulcer Scale for Healing Tool (PUSH) will be used to assess and measure change in PU status. The score on the PUSH-tool is defined by the surface area of the PU (length x width), the amount of exudate and the type of tissue in the wound bed.
  Arms: 18 residents at least one PU category III-IV in the sacral area

SUMMARY:
Pressure Ulcers are a serious and common problem for residents admitted to long-term care facilities and community care patients. They represent a major burden to patients, carers and the Healthcare system, affecting approximately 1 in 20 community patients. International guidelines recommend the use of pressure redistribution support surfaces, systematic patient repositioning and preventive skin care to prevent pressure ulcers.

It has been acknowledged that a significant proportion of pressure ulcers are avoidable. The prevalence of pressure ulcers is 1 of the 4 common harms recorded in the UK NHS Safety Thermometer, a local improvement tool for measuring, monitoring and analyzing patient harms across a range of settings, including nursing homes, community nursing and hospitals on a monthly basis.

ELIGIBILITY:
Inclusion Criteria:

* At risk of pressure ulcer development based on a Braden score ≤ 17 or pressure ulcer category III or IV
* Bedbound or chair bound
* Aged ≥ 65

Exclusion Criteria:

* Short-stay residents (expected length of stay ≤14 days)
* End of life care
* Medical contraindication for patient repositioning/turning

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-10-12 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Pressure ulcer incidence | 30 days
  Development of at least 1 Pressure ulcer category II+ during study period using European Pressure Ulcer Advisory Panel (EPUAP) classification system
Pressure ulcer healing | 30 days
  Healing of pressure ulcers category III and IV during the 30-day study period - using the Pressure Ulcer Scale for Healing Tool (PUSH)

SECONDARY OUTCOMES:
Comfort | 30 days
  perceived comfort and experiences of users of the mattress - using self-developed questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Beeckman, Phd, Principal Investigator — Study Principal Investigator
Locations (1):
- WZC Hof ter Waarbeek, Asse, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown S, Smith IL, Brown JM, Hulme C, McGinnis E, Stubbs N, Nelson EA, Muir D, Rutherford C, Walker K, Henderson V, Wilson L, Gilberts R, Collier H, Fernandez C, Hartley S, Bhogal M, Coleman S, Nixon JE. Pressure RElieving Support SUrfaces: a Randomised Evaluation 2 (PRESSURE 2): study protocol for a randomised controlled trial. Trials. 2016 Dec 20;17(1):604. doi: 10.1186/s13063-016-1703-8. PMID 27993145
- See also: Website of the research group — https://www.skintghent.be/en